CLINICAL TRIAL: NCT04613570
Title: SUrveillance of PREMalignant Stomach - Individualized Endoscopic Follow-up
Acronym: SUPREME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Portugues de Oncologia, Francisco Gentil, Porto (Other)
Responsible Party: Principal Investigator, Diogo Libânio, Principal Investigator, Instituto Portugues de Oncologia, Francisco Gentil, Porto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SUPREME
Record Dates: First submitted 2020-10-16; First posted 2020-11-03 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Atrophic Gastritis; Intestinal Metaplasia; Gastric Dysplasia; Gastric Cancer
Keywords: atrophic gastritis; gastric cancer; intestinal metaplasia; gastric dysplasia; surveillance
MeSH Terms: conditions — Gastritis, Atrophic; Stomach Neoplasms | interventions — Endoscopy, Digestive System

STUDY DESIGN:
Intervention Model Description: Patients with EGGIM > 5 or OLGA/OLGIM III/IV (premalignant stomach group - SUPREME I) will be randomized to endoscopic surveillance every one (12 to 16 months) or three years (32-40 months);
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yearly endoscopy (Experimental): Upper gastrointestinal endoscopy every year (12-16 months)
  Interventions: Diagnostic Test: Upper gastrointestinal endoscopy
- Endoscopy every 3 years (Other): Upper gastrointestinal endoscopy every three years (32-40 months)
  Interventions: Diagnostic Test: Upper gastrointestinal endoscopy

INTERVENTIONS:
Diagnostic Test: Upper gastrointestinal endoscopy — In all patient's complete gastroscopy first with White light and then with virtual chromoendoscopy will be made;
  * Suspicious lesions with dysplasia/cancer will be biopsied 1-2 fragments in a different vial; if an irregular area of mucosa (pattern C) with no clearly defined lesion then 1-2 guided biopsies fragments will be taken and sent in a different vial;
  * EGGIM (Endoscopic Grading of Gastric Intestinal Metaplasia) will be calculated according to previous description of this classification:
  * If EGGIM 0 (no endoscopically apparent IM) biopsies will be made in antrum, incisura and corpus according to Sydney-Houston protocol;
  * If EGGIM 1 or more guided biopsies of suspicious areas of IM should be made replacing the random biopsies in that particular area;
  * Antrum, incisura and corpus fragments should be sent in 3 separate vials;

SUMMARY:
Introduction: Gastric atrophy and intestinal metaplasia are the principal precursors for gastric cancer and, therefore, are considered gastric premalignant conditions. Although current guidelines recommend surveillance of individuals with these conditions, the best method for its identification and staging (histological vs endoscopy) and the best time schedule for follow-up are still controversial. Aims: To describe for the first-time patients with premalignant conditions both clinically (familial history), histologically (OLGA/OLGIM; complete/incomplete metaplasia) and endoscopically (EGGIM) using validated scales and to describe evolution of these parameters through time. To estimate prospectively the gastric cancer risk according to EGGIM stages. To define the best endoscopic surveillance follow-up for the several stages considering clinical, histological and endoscopic factors.

Methods: Multicenter study involving different gastroenterology departments from several countries. Consecutive patients older than 45 years scheduled for upper endoscopy in each of these centers will be evaluated by High-Resolution- endoscopy with virtual chromoendoscopy and EGGIM will be calculated. Guided biopsies (if areas suspicious of IM) and/or random biopsies (if no areas suspicious of IM) in antrum and corpus will be made and OLGA/OLGIM stages calculated. Patients will be evaluated in clinical consultation and database will be fulfilled. All patients will be eradicated for Helicobacter pylori infection if positive. At that occasion, all the patients with EGGIM>5 and/or OLGA III/IV and/or OLGIM III/IV will be randomized for yearly (12 to 16 months) or every three years (32-40 months) endoscopic follow-up during a period of 6 years (SUPREME I). Endoscopic observational follow-up will be scheduled for patients with EGGIM 1-4 and OLGIM I/II at 3 and 6 years (SUPREME II). For individuals with no evidence of IM (EGGIM 0 and OLGIM 0, OLGA 0-II) a follow-up endoscopy 6 years after will be proposed (SUPREME III).

DETAILED DESCRIPTION:
Introduction: Gastric atrophy and intestinal metaplasia are the principal precursors for gastric cancer and, therefore, are considered gastric premalignant conditions. Although current guidelines recommend surveillance of individuals with these conditions, the best method for its identification and staging (histological vs endoscopy) and the best time schedule for follow-up are still controversial. Aims: To describe for the first-time patients with premalignant conditions both clinically (familial history), histologically (OLGA/OLGIM; complete/incomplete metaplasia) and endoscopically (EGGIM) using validated scales and to describe evolution of these parameters through time. To estimate prospectively the gastric cancer risk according to EGGIM stages. To define the best endoscopic surveillance follow-up for the several stages considering clinical, histological and endoscopic factors.

Methods: Multicenter study involving different gastroenterology departments from several countries. Consecutive patients older than 45 years scheduled for upper endoscopy in each of these centers will be evaluated by High-Resolution-endoscopy with virtual chromoendoscopy and EGGIM will be calculated. Guided biopsies (if areas suspicious of IM) and/or random biopsies (if no areas suspicious of IM) in antrum and corpus will be made and OLGA/OLGIM stages calculated. Patients will be evaluated in clinical consultation and database will be fulfilled. All patients will be eradicated for Helicobacter pylori infection if positive. At that occasion, all the patients with EGGIM>5 and/or OLGA III/IV and/or OLGIM III/IV will be randomized for yearly (12 to 16 months) or every three years (32-40 months) endoscopic follow-up during a period of 6 years (SUPREME I). Endoscopic observational follow-up will be scheduled for patients with EGGIM 1-4 and OLGIM I/II at 3 and 6 years (SUPREME II). For individuals with no evidence of IM (EGGIM 0 and OLGIM 0, OLGA 0-II) a follow-up endoscopy 6 years after will be proposed (SUPREME III).

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for upper GI endoscopy with indication for gastric biopsies, including those with known gastric pathology (e.g. auto-immune gastritis) or premalignant conditions (e.g patients under surveillance because of atrophic gastritis);
* Age above 45 years old

Exclusion Criteria:

* History of previous gastrectomy;
* History of endoscopic resection of neoplastic lesion
* History of previous gastric dysplasia (even with no detectable lesion)
* Hereditary syndromes that increase gastric cancer risk (familial adenomatous polyposis; Lynch syndrome)
* Serious comorbidities (ASA 3 or more)
* Medication with anticoagulants

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 912 (Estimated)
Dates: Start 2021-01-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Dysplasia | 6 years
  Proportion of patients with dysplasia (low or high-grade)
Carcinoma | 6 years
  Proportion of patients with gastric adenocarcinoma

SECONDARY OUTCOMES:
Curative criteria | 6 years
  Proportion of patients with intramucosal carcinoma with low-risk criteria ("curative" criteria)
Non-curative criteria | 6 years
  Proportion of patients with submucosal, diffuse type or intramucosal carcinoma with high-risk criteria ("non-curative" criteria)
Advanced gastric cancer | 6 years
  Proportion of patients with advanced gastric cancer (without indication for endoscopic treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Pimentel-Nunes, MD PhD, Principal Investigator — Instituto Português de Oncologia do Porto, Francisco Gentil
Locations (1):
- IPO-Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/70/NCT04613570/Prot_000.pdf